CLINICAL TRIAL: NCT05822661
Title: Evaluation of the Impact of Black Seed Oil on Hemodialysis Patients
Brief Title: Impact of Black Seed Oil on Hemodialysis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 119
Record Dates: First submitted 2023-02-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-02

CONDITIONS: End Stage Renal Disease
Keywords: black seed oil; nigella sativa; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Nigella sativa oil

STUDY DESIGN:
Intervention Model Description: Drug vs placebo
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Seed Oil (Experimental): 900 mg (as two separate soft gels) twice daily for 8 weeks
  Interventions: Dietary Supplement: Black Seed Oil
- Placebo (Placebo Comparator): matched placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Black Seed Oil — Dietary supplement
  Other Names: Nigella sativa
  Arms: Black Seed Oil
Dietary Supplement: Placebo — placebo capsules same odor, color and size as the drug but without the active ingredient
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of black seed oil on endothelial dysfunction, oxidative stress and quality of life in hemodialysis patients.

DETAILED DESCRIPTION:
Evaluation of the effect of black seed oil in hemodialysis patients via:

* Evaluation of serum Endothelin-1 levels
* Evaluation of serum Malondialdehyde (MDA) levels
* Evaluation of serum Total Antioxidant Capacity (TAC) levels
* Evaluation of Quality of Life (QOL)
* Evaluation of fatigue scale

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Three to four times per week hemodialysis
* Being on hemodialysis for at least 6 months
* Ability and willingness to cooperate in the study

Exclusion Criteria:

* Pregnancy or lactation
* Cigarette smoking or substance/alcohol abuse
* Having active infectious diseases
* Receiving steroidal or nonsteroidal anti-inflammatory drugs
* Using Nigella sativa oil regularly
* Changes in treatment methods (dialysis) or medications during the supplementation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-04-23 (Estimated); Study Completion 2023-04-23 (Estimated)

PRIMARY OUTCOMES:
serum Endothelin-1 (ET-1) level | 8 weeks
  marker of endothelial dysfunction

SECONDARY OUTCOMES:
Serum malondialdehyde (MDA) and total antioxidant capacity (TAC) | 8 weeks
  markers of oxidative stress
Quality of life questionnaire | 4 weeks and 8 weeks
  using validated Arabic version SF-36 questionnaire
Fatigue severity | 4 weeks and 8 weeks
  using the Multidimensional Fatigue Inventory (MFI)

CONTACTS AND LOCATIONS:
Overall Officials: May A Shawki, PHD, Study Director — Faculty of pharmacy - Ain Shams University; Areej M Ateya, PHD, Study Director — Faculty of pharmacy - Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt